CLINICAL TRIAL: NCT00839761
Title: Efficacy of Iron Fortified Ultra Rice Compared to Supplemental Iron Drops in Infants and Young Children
Brief Title: The Use of Ultra Rice Compared to Iron Drops Consumed by Anemic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Mark Anthony Beinner, Escola de Enfermagem - UFMG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDAAA
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Anemia; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iron fortified rice group (Experimental)
  Interventions: Dietary Supplement: iron fortified rice
- iron drop group (Placebo Comparator)
  Interventions: Dietary Supplement: iron drops

INTERVENTIONS:
Dietary Supplement: iron fortified rice
  Arms: iron fortified rice group
Dietary Supplement: iron drops
  Arms: iron drop group

SUMMARY:
Background: How best to improve iron status among infants in low-income settings is of continued concern in many countries, including Brazil

Objective:

Design: In a double blind, 5-mo, home-based trial in Brazil, mildly anemic 6 - 24 month-old children (n=175) were randomly assigned to receive either Ultra Rice (URG) fortified with 23,4, mg Fe as micronized ferric pyrophosphate (MFP) and a placebo solution of iron drops, or identical non-fortified rice (CG) and a solution of iron drops. Parents were instructed on the correct dosage of iron drops and to feed their children (including whether and how much rice) as they normally would. Iron status and hemoglobin (Hb) were measured at baseline and at 5 mo.

ELIGIBILITY:
Inclusion Criteria:

* anemia

Exclusion Criteria:

* non anemic

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Before, the prevalence of ID and anemia in sample were 73.1% and 100%, respectively. At 5-mo, increases occurred in serum ferritin (SF) and hemoglobin (Hb). SF and Hb were observed in both groups. Increases in both measures were seen in the URG group. | Before and after 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Minas Gerais - UFMg, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Moretti D, Zimmermann MB, Muthayya S, Thankachan P, Lee TC, Kurpad AV, Hurrell RF. Extruded rice fortified with micronized ground ferric pyrophosphate reduces iron deficiency in Indian schoolchildren: a double-blind randomized controlled trial. Am J Clin Nutr. 2006 Oct;84(4):822-9. doi: 10.1093/ajcn/84.4.822. PMID 17023709